CLINICAL TRIAL: NCT04343833
Title: Primary Stability and PES/WES Evaluation for Immediate Implants in the Aesthetic Zone: a Clinical Double-blind Randomized Study
Brief Title: Immediate Implants in the Aesthetic Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Arturo Sánchez-Pérez, Associate professor, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2076/20018
Record Dates: First submitted 2020-04-07; First posted 2020-04-13 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Immediate Dental Implant
Keywords: Dental esthetics; Primary stability; Single-tooth restoration; Osseointegration.

STUDY DESIGN:
Intervention Model Description: A total of 20 patients, distributed in two groups with ten patient each (experimental and control) were included in this study. All patients signed a double informed consent, one for implant placement and one for their participation in the study. The study follows the Declaration of Helsinki recommendations. The Ethics Committee of the University of Murcia approved the study protocol with ID: 2076/2018.
Who Masked: Participant, Investigator
Masking Description: Double (participant, investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control with Standard dental implant (Active Comparator): Patients were treated with implants Inhex Ticare Standard (Mozo Grau, Ticare, Valladolid, Spain). The implants presented a surface treated with Reabsorbable Blast Media (RBM), conical macro-design with non-aggressive threads, internal connection, and platform switching. On the implant shoulder, the beveled design of the platform was characterized by a rounded shape of 45º.
  Interventions: Procedure: Immediate dental implants
- Test with the new implant design (Experimental): Patients were treated with Implants Inhex Quattro Ticare (Mozo Grau, Ticare, Valladolid, Spain). The implants also presented a surface treated with RBM, conical macro-design with expanded micro threads, internal connection, and platform switching.On the implant shoulder, the beveled design of the platform was characterized by a rounded shape of 45º.
  Interventions: Procedure: Immediate dental implants

INTERVENTIONS:
Procedure: Immediate dental implants — At the time of operation, the tooth was atraumatically extracted, and the implant was immediately placed following the surgical protocol recommended by the manufacturer. A temporary prosthesis was made without occlusal contact.
  Other Names: Fresh extraction sockets

SUMMARY:
The use of immediate implants in the aesthetic area is a technique widely used in modern implantology. The characteristics of the patient, the implant, and the surgical procedure used may influence the final results. The aim was to assess whether the implant design affects primary (PS) and secondary stability (SS), bone level (BL), and PES/WES evaluation.

DETAILED DESCRIPTION:
20 implants with two different designs (n=10) were immediately placed in the upper anterior maxilla with no grafting material. ISQ, BL, and PES/WES were evaluated. Results will analyze with the Wilcoxon-Mann-Whitney test (p<0.05).

The random distribution is made prior to assignment following the internet prgram https://www.random.org

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented aa vertical fracture in an upper incisor that can not be treated conservatively and ended in the extraction, and the treatment needed is a unitary implant.
* Good systemic health status (ASA I or II).
* Oral hygiene index of < 2 (Löe and Silness).
* A minimum of 2 mm of attached mucosa.
* A minimum of 8 mm of vertical bone.
* A minimum of 7 mm of bucco-lingual bone.

Exclusion Criteria:

* Traumatic or complicated incisor extraction.
* Pregnant or women in the lactation period.
* Use of any medication that contraindicates implant treatment.
* A history of alcohol or drug abuse.
* A requirement for guided bone regeneration.
* A requirement for tissue graft augmentation.
* Failure to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
Bone level | After 12 months of definitive implant load
  The bone level (BL) was determined by an intraoral digital radiograph taken parallel to the long axis of the implant.
  The distance from the implant neck to the first contact between the bone and the implant was determined. It was measured in both sides, mesial and distal, and the mean between both values was established as the BL value.
PES/WES | After 12 months of definitive implant load
  Pink Esthetic Score/White Esthetic Score [PES/WES] The parameters evaluated by this index are (1) mesial papilla, (2) distal papilla, (3) curvature of facial mucosa, (4) level of facial mucosa, and (5) root convexity/soft tissue color and texture. Each parameter range between 0 and 2. A maximum score of 10 can be obtained, considering acceptable from 6 The WES focuses specifically on the visible part of the restoration and in base on the following five parameters: (1) tooth form, (2) tooth volume/outline, (3) color (hue and value), (4) Surface texture, and (5) translucency. Each parameter is evaluated by comparison with the adjacent teeth, giving a value ranged from 0 to 2. A total score of 10 can be obtained, considering acceptable from 6

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine and Dentistry Faculty, Murcia University, Morales Meseguer Hospital, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Non-personal data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Aftr the publication of the results
Access Criteria: Any interested reseacher

REFERENCES:
- [Derived] Sanchez-Perez A, Nicolas-Silvente AI, Sanchez-Matas C, Molina-Garcia S, Navarro-Cuellar C, Romanos GE. Primary stability and PES/WES evaluation for immediate implants in the aesthetic zone: a pilot clinical double-blind randomized study. Sci Rep. 2021 Oct 8;11(1):20024. doi: 10.1038/s41598-021-99218-8. PMID 34625591